CLINICAL TRIAL: NCT05390970
Title: Platelet-Rich Plasma Injection for the Treatment of Female Stress Urinary Incontinence: A Randomized Placebo-Controlled Study
Brief Title: Platelet-Rich Plasma for Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Annah J. Vollstedt (Other)
Responsible Party: Sponsor-Investigator, Annah J. Vollstedt, Principle investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202112270
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Urinary Incontinence,Stress; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet-rich Plasma (Experimental): These subjects will have the active PRP injected into their anterior vaginal wall.
  Interventions: Procedure: Platelet-rich plasma injection
- Placebo (saline) (Placebo Comparator): These subjects will have a saline placebo injected into the anterior vaginal wall.
  Interventions: Procedure: Platelet-rich plasma injection

INTERVENTIONS:
Procedure: Platelet-rich plasma injection — Injection of autologous platelet-rich plasma into the anterior vaginal wall

SUMMARY:
The aim of this randomized controlled trial study is to evaluate the efficacy and safety of platelet-rich plasma (PRP) in the treatment of female stress urinary incontinence (SUI), compared to placebo. Subjects will undergo an injection of PRP (or injectable saline placebo) into the anterior vaginal wall in the office. Primary outcomes will include a negative urinary stress test plus improvement with the Patient Global Impression of Improvement (PGI-I) at 6-months. Secondary outcomes will include the Female Sexual Function Index (FSFI), the Incontinence Quality of life (I-QOL), Questionnaire for Urinary Incontinence Diagnosis (QUID), and the visual analog scale for pain.

DETAILED DESCRIPTION:
Platelet-rich plasma (PRP) is an autologous solution of human plasma with a high concentration of platelets. While the preparation and injection of PRP is not a new technology, it has not been well-studied in the field of urogynecology. Small case series have suggested PRP may be used in the treatment of stress urinary incontinence (SUI). The aim of this randomized controlled trial study is to evaluate the efficacy and safety of PRP in the treatment of female SUI, compared to placebo. Adult females with SUI or with stress-predominant mixed urinary incontinence will be eligible. Subjects will undergo an injection of PRP (or injectable saline) into the anterior vaginal wall in the office. At baseline and at time points of 1, 3, and 6 months, subjects will complete the validated questionnaires. A pelvic exam with a stress test will be performed by a blinded provider at the 3 and 6-month visits. Primary outcomes will include a negative urinary stress test plus improvement with the Patient Global Impression of Improvement (PGI-I) at 6-months. Secondary outcomes will include the Female Sexual Function Index (FSFI), the Incontinence Quality of life (I-QOL), Questionnaire for Urinary Incontinence Diagnosis (QUID), and the visual analog scale for pain.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years or older
2. Pure or stress-predominant urinary incontinence with the Medical, Epidemiologic, and Social Aspects of Aging questionnaire (MESA) stress incontinence symptom score greater than MESA urge incontinence symptom score
3. Observation of leakage by provocative stress test at bladder volume £ 300 mL [15]
4. Post void residual < 150 mL

Exclusion Criteria:

1. Currently pregnant or trying to conceive
2. Currently breastfeeding
3. Interstitial cystitis
4. Urgency urinary incontinence predominance or currently being treated for overactive bladder with medication, percutaneous tibial nerve stimulation, bladder chemodenervation, or sacral neuromodulation
5. Currently being treated for a sexually transmitted disease
6. Pelvic organ prolapse greater than stage 2 according to the Pelvic Organ Prolapse Quantification System
7. Periurethral mass
8. Active gynecologic, urologic or colorectal cancer
9. History of pelvic radiation
10. Psychological disorder making the patient unable to provide consent
11. Undiagnosed abnormal uterine bleeding
12. Genitourinary fistula
13. Prior SUI surgery
14. Use of anti-platelet or anti-coagulant medication
15. Regular use of non-steroidal anti-inflammatorie

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from May 2022 to April 2023 in a large academic medical institution.
Period: Overall Study
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Started | 25 | 25
Completed | 24 | 23
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Plasma | Placebo (Saline) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [40 to 55] | 45 [39 to 53] | 47 [39 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative Urinary Stress Test (no Leakage Noted on Examination During Cough or Valsalva Maneuvers at a Standardized Bladder Volume of 300 mL)
Description: Negative urinary stress test (no leakage noted on examination during cough or Valsalva maneuvers at a standardized bladder volume of 300 mL
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 24 | 25
Participants | 15 | 16

2. Primary Outcome: Subjective Outcome With Improvement in the Patient Global Impression of Improvement (PGI-I), With Positive Response Defined as "Very Much Better" (1) or "Much Better" (2)
Description: Answered "very much better" or "much better" on the Patient Global Impression of Improvement (PGI-I)
Time Frame: 6-months
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 25 | 24
Participants | 4 | 1

3. Secondary Outcome: Female Sexual Function Index (FSFI) Scores
Description: 6-months FSFI score in the PRP group versus the saline group. Score range is 0-36, the higher the value the greater the level of sexual functioning. Scale ranges from 0 "No sexual activity", 1 "Almost never or never" to 5 "Almost always or always" OR 0 "No sexual activity", 1 "Extremely difficult or impossible" to 5 "Not difficult".
Time Frame: 6-months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 25 | 25
score on a scale | 27 [22 to 31] | 25 [17 to 31]

4. Secondary Outcome: Incontinence-Quality of Life (I-QOL) Scores
Description: How the subject's quality of life is different related to urinary leakage after the procedure based on their I-QOL score. Score ranges from 22-110, the higher the score the better their quality of life. Scale goes from 1 "Extremely' to 5 "Not at all".
Time Frame: 6-months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 25 | 23
score on a scale | 87 [75 to 102] | 88 [62 to 94]

5. Secondary Outcome: Questionnaire for Urinary Incontinence Diagnosis (QUID)
Description: How severe the urinary leakage is after the procedure based on the QUID score. Score ranges from 0-30. Scale ranges from 0 "None of the time" to 5 "All of the time".
Time Frame: 6-months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 25 | 23
score on a scale | 10.0 [7.0 to 13.0] | 10.0 [6.0 to 14.5]

6. Secondary Outcome: Perception of Monetary Value
Description: How much money the subject would be willing to pay for the procedure; this was a free text question
Time Frame: 6-months
Measure: Median (Inter-Quartile Range); unit: US dollars
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 25 | 25
US dollars | 100 [50 to 200] | 50 [0 to 100]

7. Secondary Outcome: Visual Analog Scale (VAS) for Patient Pain/Discomfort
Description: How painful the procedure itself is from 0 to 10 with 0 being no pain and 10 being "pain as bad as it could be"
Time Frame: after injection
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 25 | 25
units on a scale | 2.25 (1.45) | 2.87 (2.07)

8. Secondary Outcome: Visual Analog Scale (VAS) for Procedure Difficulty (by Provider)
Description: how difficult the procedure is for the patient on a scale from 0 to 10 with 0 being not difficult at all and 10 being the most difficult procedure to perform
Time Frame: after injection
Measure: Number; unit: units on a scale
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
Number analyzed (Participants) | 25 | 25
units on a scale | 2 | 2.54

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 6 months after the procedure was performed.
Description: All participants were at risk for serious adverse events
Arm/Group | Platelet-rich Plasma | Placebo (Saline)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 23/25 | 23/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platelet-rich Plasma (N=25) | Placebo (Saline) (N=25)
Vaginal spotting (Surgical and medical procedures) | 6 (6) | 6 (6)
Heavy Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Burning with urination (Renal and urinary disorders) | 1 (1) | 1 (1)
Blood in urine (Renal and urinary disorders) | 4 (4) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 4 (4)
Vaginal discomfort (General disorders) | 7 (7) | 9 (9)
vaginal pain (General disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT05390970/Prot_SAP_000.pdf